CLINICAL TRIAL: NCT05397392
Title: Research on Optimal Diagnosis and Treatment of Cardiorenal Syndrome
Acronym: ODT-CRS
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: KY20220425-02
Record Dates: First submitted 2022-05-26; First posted 2022-05-31 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-04

CONDITIONS: Heart Failure; Kidney Diseases; Kidney Injury; Heart Valve Diseases; Dialysis; Complications; Coronary Heart Disease
MeSH Terms: conditions — Heart Failure; Kidney Diseases; Heart Valve Diseases; Coronary Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- acute kidney injury: Acute kidney injury caused by heart disease or cardiac dysfunction due to acute renal damage
  Interventions: Other: guideline recommended routine treatment
- chornic kidney disease: Chornic kidney injury caused by heart disease or cardiac dysfunction due to chronic kidney disease
  Interventions: Other: guideline recommended routine treatment

INTERVENTIONS:
Other: guideline recommended routine treatment

SUMMARY:
To estimate the characteristics, pathogenesis, risk factors and intervention measures for different stages of heart and kidney diseases, and to optimize the curative effects of different treatment schemes

DETAILED DESCRIPTION:
Cardiorenal syndrome is a clinical syndrome caused by acute or chronic injury of one of the heart and kidney resulting to acute or chronic dysfunction of the other organ. In recent years, the morbidity of cardiorenal syndrome has increased rapidly in China. Its condition is complex and difficult to treat. Due to the lack of studies specifically targeting the cardiorenal syndrome population, there is no systematic in-depth understanding of the pathogenesis and risk factors of this kind of disease. In clinic, the course of various types of cardiorenal syndrome is complex and difficult to be summarized into a specific type. Therefore, we intend to conduct a clinical systematic observation and research on such patients so as to optimize a more reasonable treatment scheme.

ELIGIBILITY:
Inclusion Criteria:

Patients meet the diagnosis of various types of cardiorenal syndrome according to the classification standards of various types formulated by KDIGO and ADQI expert consensus. Different syndromes were identified and classified into five subtypes. Acute CRS (type 1): acute worsening of heart function (AHF-ACS) leading to kidney injury and/or dysfunction. Chronic cardio-renal syndrome (type 2): chronic abnormalities in heart function (CHF-CHD) leading to kidney injury and/or dysfunction. Acute reno-cardiac syndrome (type 3): acute worsening of kidney function (AKI) leading to heart injury and/or dysfunction. Chronic reno-cardiac syndrome (type 4): chronic kidney disease leading to heart injury, disease, and/or dysfunction. Secondary CRS (type 5): systemic conditions leading to simultaneous injury and/or dysfunction of heart and kidney.

Exclusion Criteria:

Pregnant or breastfeeding women; Female patients with recent birth plans; Patients who cannot follow up on medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients from a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Hospitalization due to worsening of renal or cardiac function | 1 year
  eGFR continuously decreased by more than 25% within one year; NYHA cardiac function class III or above requires intravenous pharmacological agents; deterioration of cardiac or kidney function requiring dialysis
All-cause deaths | 1 year
  Deaths due to disease progression

SECONDARY OUTCOMES:
End-stage renal disease requires maintenance dialysis | 1 year
  eGFR<15ml/min, combined with one of the following conditions: 1. Uremia symptoms that cannot be alleviated by limiting protein intake; 2. Hyperkalemia that is difficult to correct; 3. Progressive metabolic acidosis that is difficult to control; 4. Uncontrollable water and sodium retention, combined with congestive heart failure or acute pulmonary edema; 5. Uremic pericarditis; 6. Uremic encephalopathy and progressive neuropathy.
Acute kidney injury | 1 year
  increase in Scr ≥0.3 mg/dL (26.5 μmol/L) within 48 h, or increase in Scr ≥1.5 times baseline in 7 days, or urine volume <0.5 mL/kg/h for 6 h.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing, China